CLINICAL TRIAL: NCT02503800
Title: The Significance of Blood-tryptase Levels and c-Kit Mutation in the Evaluation of Prognosis and Adverse Reactions in Subjects Undergoing Venom Immunotherapy for Insect Allergy
Brief Title: The Significance of Blood-tryptase and c-Kit Mutation in Insect Venom Immunotherapy
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, alon hershko, Chairman, Department of Medicine B, Meir Medical Center
Other Study IDs: MMC150100-15CTIL
Record Dates: First submitted 2015-07-16; First posted 2015-07-21 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Hypersensitivity, Immediate; Insect Bites and Stings; Mastocytosis
MeSH Terms: conditions — Hypersensitivity, Immediate; Insect Bites and Stings; Mastocytosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen will include 5 ml of venous whole blood drawn for measurement of serum tryptase and leukocyte c-Kit mutation.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- subjects undergoing venom immunotherapy: The study group will include all the subjects receiving routine venom immunotherapy at the Meir Medical Center Allergy Clinic.

SUMMARY:
The investigators wish to evaluate the association between tryptase values as well as c-Kit mutation and adverse effects in the course of immunotherapy. The investigators also intend to assess the effect of immunotherapy on tryptase levels.

DETAILED DESCRIPTION:
According to the presently available reports there is an association between systemic allergic responses to hymenoptera venom and elevated tryptase levels or c-Kit mutation. The presence of these findings may imply the existence of mast cell activation syndrome or mastocytosis. Therefore, baseline tryptase evaluation has become standard evaluation in patients with systemic responses. Meir Medical Center is the only hospital in Israel in which tryptase can be measured. Consequently, the Meir Clinic has accumulated considerable data with regards to tryptase levels in subjects with allergy to hymenoptera venom. The investigators wish to evaluate the association between tryptase values as well as c-Kit mutation and adverse effects in the course of immunotherapy. The investigators also intend to assess the effect of immunotherapy on tryptase levels.

ELIGIBILITY:
Inclusion Criteria:

* history of systemic response to hymenoptera sting.
* subject under current or planned venom immunotherapy.

Exclusion Criteria:

* previously diagnosed mast cell disorder

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population will include all the subjects undergoing venom immunotherapy at the Clinic of Allergy and Clinical Immunology, Meir Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2015-08; Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
The association between tryptase values/c-Kit mutation and immunotherapy adverse events will be evaluated using blood sample analysis and patient medical records. | up to 12 months

SECONDARY OUTCOMES:
The association between tryptase values/c-Kit mutation and severity of index sting event will be evaluated using blood sample analysis and patient medical records. | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alon Y Hershko, MD, PhD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Cichocka-Jarosz E, Sanak M, Szczeklik A, Brzyski P, Pietrzyk JJ. Impact of Hymenoptera venom allergy and the effects of specific venom immunotherapy on mast cell metabolites in sensitized children. Ann Agric Environ Med. 2014;21(2):294-301. doi: 10.5604/1232-1966.1108594. PMID 24959779
- [Background] Niedoszytko M, de Monchy J, van Doormaal JJ, Jassem E, Oude Elberink JN. Mastocytosis and insect venom allergy: diagnosis, safety and efficacy of venom immunotherapy. Allergy. 2009 Sep;64(9):1237-45. doi: 10.1111/j.1398-9995.2009.02118.x. Epub 2009 Jul 21. PMID 19627278
- [Result] Zanotti R, Lombardo C, Passalacqua G, Caimmi C, Bonifacio M, De Matteis G, Perbellini O, Rossini M, Schena D, Busa M, Marcotulli MC, Bilo MB, Franchini M, Marchi G, Simioni L, Bonadonna P. Clonal mast cell disorders in patients with severe Hymenoptera venom allergy and normal serum tryptase levels. J Allergy Clin Immunol. 2015 Jul;136(1):135-9. doi: 10.1016/j.jaci.2014.11.035. Epub 2015 Jan 17. PMID 25605272